CLINICAL TRIAL: NCT06362304
Title: Application of 99mTc-CNDG SPECT/CT Imaging in the Diagnosis of Brain Tumors
Brief Title: 99mTc-CNDG SPECT/CT in Brain Tumors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024-DG-01
Record Dates: First submitted 2024-04-09; First posted 2024-04-12 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Intracranial Tumor
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intracranial tumor (Experimental)
  Interventions: Diagnostic Test: 99mTc-CNDG SPECT/CT

INTERVENTIONS:
Diagnostic Test: 99mTc-CNDG SPECT/CT — FDG-PET and 99mTc-CNDG will be performed within 2 weeks before surgery.

SUMMARY:
The goal of this clinical trial is to evaluate the value of 99mTc-CNDG for diagnosis of brain tumors by comparing it with 18F-FDG-PET. The main questions it aims to answer are:

1. What is the diagnostic consistency between 99mTc-CNDG and 18F-FDG?
2. What is the correlation between the SUVmax value of 99mTc-CNDG and tumor type?

Participants will:

Receive18F-FDG-PET and 99mTc-CNDG examination within 2 weeks before surgery. Obtain pathological diagnosis by surgery or biopsy as the gold standard.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical diagnosis of brain tumor;
* Be at least 18 years old;
* The final pathological results could be obtained by surgery or biopsy;
* Informed consent and the ability to be followed up;
* Those who did not meet the exclusion criteria.

Exclusion Criteria:

* Insulin-dependent diabetes mellitus or fasting blood glucose >7 mmol/L before 99mTc-CNDG injection;
* Severe liver or kidney disease (serum creatinine level >3.0mg/dL or any liver enzyme level ≥ 5 times the upper limit of normal);
* Severe hypersensitivity or hypersensitivity to radiocontrast agents;
* Claustrophobia (inability to undergo SPECT/CT or PET/CT scans);
* Patients receiving radiotherapy and chemotherapy;
* Being pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-20 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
SUVmax | 1month
  1. Diagnostic consistency evaluation of 99mTc-CNDG and 18F-FDG; 2.Correlation of SUV value of 99mTc-CNDGwith tumor type

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No